CLINICAL TRIAL: NCT04800705
Title: Levels of Zinc (Zn), Copper (Cu), Calcium (Ca), Iron (Fe), Manganese (Mn), Selenium (Se), Strontium (Sr), Aluminium (Al), Antimonium (Sb), Phosphorus (P), Magnesium (Mg), Sodium (Na), Potassium (K), Barium (Ba) and Thallium (Tl) in Idiopathic Premature Ovarian Failure
Brief Title: Levels of Selected Macroelements in Premature Ovarian Insufficiency
Acronym: POİ&MACROs
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cengiz Gokcek Women's and Children's Hospital (Other)
Collaborators: The Scientific Research Project Fund of Yozgat Bozok University (Unknown)
Responsible Party: Principal Investigator, Ali Ovayolu, Principal Investigator, Cengiz Gokcek Women's and Children's Hospital
Other Study IDs: CengizGWCH23
Record Dates: First submitted 2021-03-11; First posted 2021-03-16 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Premature Ovarian Failure
MeSH Terms: conditions — Primary Ovarian Insufficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Premature ovarian insufficiency (POI): POI is a clinical syndrome defined by loss of ovarian activity before the age of 40 years. POI is characterized by menstrual disturbance (amenorrhea or oligomenorrhea) with raised gonadotropins and low estradiol.
  Interventions: Other: ultrasound assessment
- Control group: The study population will be consisted of 70 women with POI as the study group and 70 patients with normal healthy women as the control group. A volunteer group of healthy women who will be visited the gynaecology clinic for routine examinations and women who will be admitted for pre-pregnancy tests will be invited randomly to this research as a control group.
  Interventions: Other: ultrasound assessment

INTERVENTIONS:
Other: ultrasound assessment — Zinc (Zn), copper (Cu), calcium (Ca), iron (Fe), manganese (Mn), selenium (Se), strontium (Sr), aluminum (Al), antimonium (Sb), phosphorus (P), magnesium (Mg), sodium (Na), potassium (K), barium (Ba) and thallium (Tl) measurements (µg/L,mean±SD)
  Other Names: elements concentrations measurements

SUMMARY:
Aim: To evaluate plasma zinc (Zn), copper (Cu), calcium (Ca), iron (Fe), manganese (Mn), selenium (Se), strontium (Sr), aluminum (Al), antimonium (Sb), phosphorus (P), magnesium (Mg), sodium (Na), potassium (K), barium (Ba) and thallium (Tl) levels in women with premature ovarian insufficiency (POI) and to compare the results with those of healthy subjects.

Methods: This prospective study will be included 70 women with idiopathic premature ovarian insufficiency and 70 controls. The blood/urine/hair for analyses will be obtained at the early follicular phase of the menstrual cycle and plasma zinc (Zn), copper (Cu), calcium (Ca), iron (Fe), manganese (Mn), selenium (Se), strontium (Sr), aluminum (Al), antimonium (Sb), phosphorus (P), magnesium (Mg), sodium (Na), potassium (K), barium (Ba) and thallium (Tl) levels will be measured using inductively coupled plasma-mass spectrometry.

DETAILED DESCRIPTION:
This will be an observational prospective cohort study conducted at Obstetrics and Gynecology Department of Cengiz Gokcek Obstetrics and Children's Hospital between January 2020 and September 2021. The authors will be recruited 70 subjects with idiopathic POI, and 70 healthy patients were selected for the control group. All patients will be given their oral and written informed consent before their inclusion in the study. The protocol was approved by the Ethics Committee for Clinical Research of Gaziantep University (Reference number: 2021/343). The study strictly will be adhered to the principles of the Declaration of Helsinki.

Women between the ages of 18-39 will be included. A volunteer group of healthy women who will be visited the gynecology clinic for routine examinations and women who will be admitted for pre-pregnancy tests will be invited randomly to this research as a control group. Healthy women, who will be returned during their early follicular phase of the menstrual cycle, will be recruited as the control group subjects. The exclusion criteria will be as follows: women with evidence for karyotypic, metabolic, toxic, or iatrogenic cause of the ovarian insufficiency and any women who use any medication for POI treatment. At enrollment, for both groups, the authors will be collected data about age, height, weight, BMI, age of menarche, obstetrics history, history of smoking, regular exercise and family history of POI. At enrolment, all patients will be underwent vaginal ultrasonography for the assessment of antral follicle count (AFC) and venous blood sample from the antecubital veins for measuring plasma concentration of zinc (Zn), copper (Cu), calcium (Ca), iron (Fe), manganese (Mn), selenium (Se), strontium (Sr), aluminum (Al), antimonium (Sb), phosphorus (P), magnesium (Mg), sodium (Na), potassium (K), barium (Ba) and thallium (Tl), Follicle-stimulating hormone (FSH), E2, anti-mullerian hormone (AMH) and complete blood count (CBC). In control subjects, venous blood samples and AFC will be collected during the early follicular phase of the menstrual cycle. Urine and hair samples will be collected at the same time. The plasma and urine samples will be stored in aliquots at -80°C prior to the analyses of zinc (Zn), copper (Cu), calcium (Ca), iron (Fe), manganese (Mn), selenium (Se), strontium (Sr), aluminum (Al), antimonium (Sb), phosphorus (P), magnesium (Mg), sodium (Na), potassium (K), barium (Ba) and thallium (Tl). Hair samples will be stored in envelopes at room temperature. The plasma/urine/hair zinc (Zn), copper (Cu), calcium (Ca), iron (Fe), manganese (Mn), selenium (Se), strontium (Sr), aluminum (Al), antimonium (Sb), phosphorus (P), magnesium (Mg), sodium (Na), potassium (K), barium (Ba) and thallium (Tl) level will be measured using inductively coupled plasma-mass spectrometry. Then, this study will be determined plasma/urine/hair zinc (Zn), copper (Cu), calcium (Ca), iron (Fe), manganese (Mn), selenium (Se), strontium (Sr), aluminum (Al), antimonium (Sb), phosphorus (P), magnesium (Mg), sodium (Na), potassium (K), barium (Ba) and thallium (Tl) levels in women with POI (n=70) compared to those of volunteer healthy women (n=70). Then, these macroelements levels will be compared in both groups.

ELIGIBILITY:
Inclusion Criteria:

* women with idiopathic POI
* Healthy women

Exclusion Criteria:

1. women with any systemic condition (such as chronic hypertension, renal disease)
2. history of using any medication
3. drug user
4. history/presence of malignancy
5. history of Radiotherapy/chemotherapy
6. polycystic ovary syndrome
7. endometriosis
8. Patients whose chromosome analysis result is not normal
9. history of ovarian surgery
10. Ovarian cysts/mass
11. pregnancy
12. lactation

Ages: 18 Years to 39 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — POI is a clinical syndrome defined by loss of ovarian activity before the age of 40 years. POI is characterized by menstrual disturbance (amenorrhea or oligomenorrhea) with raised gonadotrophins and low estradiol. It is estimated to affect 1% of women under the age of 40, 0.1% under 30 and 0.01% under 20.
Study Population: The investigators consecutively will be recruited 70 subjects with POI, and 70 healthy women will be selected for the control group.
Sampling Method: Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2021-03-15 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
macroelements levels in the idiopathic POI group and control group | 1 week
  The primary outcome in these analyses will compare zinc (Zn), copper (Cu), calcium (Ca), iron (Fe), manganese (Mn), selenium (Se), strontium (Sr), aluminium (Al), antimonium (Sb), phosphorus (P), magnesium (Mg), sodium (Na), potassium (K), barium (Ba) and thallium (Tl) levels (µg/L,mean±SD) in the idiopathic POI group and control group.

CONTACTS AND LOCATIONS:
Locations (1):
- Cengiz Gokcek Women's and Children's Hospital., Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] European Society for Human Reproduction and Embryology (ESHRE) Guideline Group on POI; Webber L, Davies M, Anderson R, Bartlett J, Braat D, Cartwright B, Cifkova R, de Muinck Keizer-Schrama S, Hogervorst E, Janse F, Liao L, Vlaisavljevic V, Zillikens C, Vermeulen N. ESHRE Guideline: management of women with premature ovarian insufficiency. Hum Reprod. 2016 May;31(5):926-37. doi: 10.1093/humrep/dew027. Epub 2016 Mar 22. PMID 27008889
- [Result] Maclaran K, Horner E, Panay N. Premature ovarian failure: long-term sequelae. Menopause Int. 2010 Mar;16(1):38-41. doi: 10.1258/mi.2010.010014. No abstract available. PMID 20424285
- [Result] Verma P, K Sharma A, Shankar H, Sharma A, Rao DN. Role of Trace Elements, Oxidative Stress and Immune System: a Triad in Premature Ovarian Failure. Biol Trace Elem Res. 2018 Aug;184(2):325-333. doi: 10.1007/s12011-017-1197-6. Epub 2017 Nov 27. PMID 29181820
- [Result] Ekiz Yilmaz T, Tasdemir M, Kaya M, Arican N, Ahishali B. The effects of magnesium sulfate on cyclophosphamide-induced ovarian damage: Folliculogenesis. Acta Histochem. 2020 Feb;122(2):151470. doi: 10.1016/j.acthis.2019.151470. Epub 2019 Dec 4. PMID 31812447

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-12): https://cdn.clinicaltrials.gov/large-docs/05/NCT04800705/Prot_SAP_000.pdf